CLINICAL TRIAL: NCT02256267
Title: Effects of CYP3A Induction by Rifampin on the Pharmacokinetics of LY2835219 and Its Metabolites in Healthy Subjects
Brief Title: A Study of LY2835219 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15174; I3Y-MC-JPBF (Other: Eli Lilly and Company)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2014-10-01; First posted 2014-10-03 (Estimated); Results first posted 2018-08-02 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2018-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — abemaciclib; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2835219 (Experimental): Single oral dose of LY2835219
  Interventions: Drug: LY2835219
- LY2835219 + Rifampin (Experimental): Single oral dose of LY2835219 with rifampin orally, once daily for 14 days
  Interventions: Drug: LY2835219; Drug: Rifampin

INTERVENTIONS:
Drug: LY2835219 — Administered orally
  Other Names: abemaciclib
Drug: Rifampin — Administered orally
  Arms: LY2835219 + Rifampin

SUMMARY:
The aim of this two-period study is to compare how much of the study drug gets into the blood stream when it is given as a single oral dose and when it is given as a single oral dose in combination with rifampin (a Food and Drug Administration [FDA] approved antibiotic that is used to treat tuberculosis, a bacterial infection that mainly affects the lungs, and other infections). Each participant will complete both study periods.

The study will last about 34 days. Screening is required within 28 days before study drug is given.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy sterile males or surgically sterile females or postmenopausal females
* Have a body mass index (BMI) of 18 to 32 kilogram per meter square (kg/m^2)

Exclusion Criteria:

* Have participated in a clinical trial involving investigational product within the last 30 days
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal blood pressure
* Show evidence of human immunodeficiency virus (HIV), hepatitis B or hepatitis C
* Have donated blood of more than 500 milliliters (mL) within the last month
* Have used or intend to use over-the-counter or prescription medication including herbal medications within 7 days prior to dosing or during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is an open-label, 2-period, fixed-sequence study
Groups:
- LY2835219 Then LY2835219 + Rifampin: Single oral dose of 200 milligrams (mg) LY2835219 on Day 1 in Period 1. Once daily (QD) doses of 600 mg of Rifampin for 6 days (Day 1 through Day 6) in Period 2.Single oral dose of 200 mg of LY2835219 with 600 mg Rifampin orally, QD on Day 7 in Period 2. QD doses of 600 mg Rifampin was continued for 7 days in Period 2 after coadministration with LY2835219 dose.
Period: Period 1 (Day 1; Day 2 to Day 9 Washout)
Arm/Group | LY2835219 Then LY2835219 + Rifampin
Started | 24
Received at Least 1 Dose of LY2835219 | 24
Completed | 23
Not Completed | 1
Not completed — Adverse Event | 1
Period: Period 2 (Day 1 to Day 6)
Arm/Group | LY2835219 Then LY2835219 + Rifampin
Started | 23
Received at Least 1 Dose of Rifampin | 23
Completed | 23
Not Completed | 0
Period: Period 2 (Day 7 to Day 14)
Arm/Group | LY2835219 Then LY2835219 + Rifampin
Started | 23
Received LY2835219 + Rifampin | 23
Completed | 22
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- LY2835219 Alone, Then Rifampin, Then LY2835219 + Rifampin: Single oral dose of 200 mg LY2835219 on Day 1 in Period 1. Day 2 through Day 9 in Period 1 is washout. QD doses of 600 mg of Rifampin for 6 days (Day 1 through Day 6) in Period 2.
Arm/Group | LY2835219 Alone, Then Rifampin, Then LY2835219 + Rifampin
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 15
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY2835219
Time Frame: Period 1: Day 1- Predose,1, 2, 4, 6, 8, 10 hours, Days 2-9: 24, 48, 72, 96, 120, 144, 168, and 192 hours; Period 2: Day 7- Predose,1, 2, 4, 6, 8, 10 hours, Days 8-15: 24, 48, 72, 96, 120, 144, 168, 192 hours
Population: All participants who received at least 1 dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/ml)
Groups:
- 200 mg LY2835219: Single oral dose of 200 mg LY2835219
- 200 mg LY2835219 + 600 mg Rifampin: Single oral dose of 200 mg of LY2835219 with 600 mg rifampin orally, QD for 14 days
Arm/Group | 200 mg LY2835219 | 200 mg LY2835219 + 600 mg Rifampin
Number analyzed (Participants) | 24 | 21
nanogram per milliliter (ng/ml) | 134 (45) | 10.5 (58)
Statistical Analysis 1: Comparison: 200 mg LY2835219 vs 200 mg LY2835219 + 600 mg Rifampin; Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 0.0771, 90% CI 2-sided [0.0671 to 0.0886]

2. Primary Outcome: PK: Area Under the Concentration Time Curve AUC(0-∞) of LY2835219
Time Frame: as for outcome 1
Population: All participants who received at least 1 dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram x hour per mL (ng x h/mL)
Arm/Group | 200 mg LY2835219 | 200 mg LY2835219 + 600 mg Rifampin
Number analyzed (Participants) | 24 | 14
nanogram x hour per mL (ng x h/mL) | 4570 (53) | 229 (48)
Statistical Analysis 1: Comparison: 200 mg LY2835219 vs 200 mg LY2835219 + 600 mg Rifampin; Test type: Superiority or Other; Ratio of Geometric Least Squares Means = 0.0467, 90% CI 2-sided [0.0376 to 0.0581]

ADVERSE EVENTS:
Groups:
- LY2835219: Single oral dose of 200 mg LY2835219 Day 1, period 1.
- Rifampin: Single oral, QD doses of 600 mg of Rifampin for 6 days Day 1 to Day 6 in period 2
- LY2835219 + Rifampin: Single oral dose of 200 mg of LY2835219 with 600 mg rifampin orally, QD on Day 7 of period 2.
Arm/Group | LY2835219 | Rifampin | LY2835219 + Rifampin
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 1/23
Other Adverse Events (participants affected / at risk) | 8/24 | 2/23 | 4/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2835219 (N=24) | Rifampin (N=23) | LY2835219 + Rifampin (N=23)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2835219 (N=24) | Rifampin (N=23) | LY2835219 + Rifampin (N=23)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Research Organization (CRO) and its third party contractors shall not publish, discuss or release data emanating from a Study without Lilly's express written permission.